CLINICAL TRIAL: NCT01815242
Title: Adjuvant Dynamic Marker-Adjusted Personalized Therapy Trial Optimizing Risk Assessment and Therapy Response Prediction in Early Breast Cancer - Triple Negative Breast Cancer
Acronym: ADAPT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM06 / ADAPT TN
Record Dates: First submitted 2013-03-18; First posted 2013-03-21 (Estimated); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Experimental): nab-Paclitaxel + gemcitabine
  Interventions: Drug: nab-Paclitaxel; Drug: Gemcitabine
- Arm B (Experimental): nab-Paclitaxel + carboplatin
  Interventions: Drug: nab-Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: nab-Paclitaxel
Drug: Gemcitabine
  Arms: Arm A
Drug: Carboplatin
  Arms: Arm B

SUMMARY:
The trial will evaluate the optimal treatment with nab-paclitaxel in combination with either carboplatin or gemcitabine for patients with triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria

* Female patients, age at diagnosis 18 years and above (consider patients at 70 years and above for ADAPT Elderly)
* Histologically confirmed unilateral primary invasive carcinoma of the breast
* Clinical T1 - T4 (except inflammatory breast cancer)
* All clinical N (cN)
* No clinical evidence for distant metastasis (M0)
* Known HR status and HER2 status (local pathology)
* Tumor block available for central pathology review
* Performance Status ECOG < 1 or KI > 80 %
* Negative pregnancy test (urine or serum) within 7 days prior to start of induction treatment in premenopausal patients
* Written informed consent prior to beginning specific protocol procedures, including expected cooperation of the patients for the treatment and follow-up, must be obtained and documented according to the local regulatory requirements
* The patient must be accessible for treatment and follow-up

Additional Inclusion Criteria for patients receiving chemotherapy:

* Laboratory requirements for patients receiving neoadjuvant chemotherapy (within 14 days prior to induction treatment):

  * Leucocytes >= 3.5 10^9/L
  * Platelets >= 100 10^9/L
  * Hemoglobin >= 10 g/dL
  * Total bilirubin <= 1 x ULN
  * ASAT (SGOT) and ALAT (SGPT) <= 2.5 x UNL
  * Creatinine <= 175 µmol/L (2 mg/dl)
* LVEF within normal limits of each institution measured by echocardiography and normal ECG (within 42 days prior to induction treatment)

Exclusion Criteria:

* Known hypersensitivity reaction to the compounds or incorporated substances
* Prior malignancy with a disease-free survival of < 10 years, except curatively treated basalioma of the skin or pTis of the cervix uteri
* Non-operable breast cancer including inflammatory breast cancer
* Previous or concurrent treatment with cytotoxic agents for any reason after consultation with the sponsor
* Concurrent treatment with other experimental drugs. Participation in another interventional clinical trial with or without any investigational not marketed drug within 30 days prior to study entry
* Male breast cancer
* Concurrent pregnancy; patients of childbearing potential must implement a highly effective (less than 1% failure rate) non-hormonal contraceptive measures during the study treatment
* Breast feeding woman
* Sequential breast cancer
* Reasons indicating risk of poor compliance
* Patients not able to consent

Additional Exclusion Criteria for patients receiving chemotherapy:

* Known polyneuropathy ≥ grade 2
* Severe and relevant co-morbidity that would interact with the application of cytotoxic agents or the participation in the study including acute cystitis and ischuria and chronic kidney disease
* Uncompensated cardiac function
* Inadequate organ function including:

  * Leucocytes < 3.5 x 10^9/l
  * Platelets < 100 x 10^9/l
  * Bilirubin above normal limits
  * Alkaline phosphatase > 5 x UNL
  * ASAT and/or ALAT associated with AP > 2.5 x UNL

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Comparison: pCR in nab-paclitaxel/carboplatin vs. nab-paclitaxel/gemcitabine | After 12 weeks of therapy
  pCR will be measured after 12 weeks of randomized treatment.
Comparison: pCR in responders vs. non-responders | After 12 weeks of therapy
  pCR will be measured after 12 weeks of randomized treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Harbeck, Prof. Dr., Principal Investigator — Breast Center of the University of Munich (LMU), Universitätsfrauenklinik Großhadern, Munich, Germany; Ulrike Nitz, Prof. Dr., Study Chair — Ev. Krankenhaus Bethesda Brustzentrum Niederrhein, Mönchengladbach, Germany
Locations (1):
- Ev. Krankenhaus Bethesda Brustzentrum Niederrhein, Mönchengladbach, Germany, Mönchengladbach, Germany

REFERENCES:
- [Background] Hofmann D, Nitz U, Gluz O, Kates RE, Schinkoethe T, Staib P, Harbeck N. WSG ADAPT - adjuvant dynamic marker-adjusted personalized therapy trial optimizing risk assessment and therapy response prediction in early breast cancer: study protocol for a prospective, multi-center, controlled, non-blinded, randomized, investigator initiated phase II/III trial. Trials. 2013 Aug 19;14:261. doi: 10.1186/1745-6215-14-261. PMID 23958221
- [Derived] Korbie D, Stirzaker C, Gluz O, Zu Eulenburg C, Nitz U, Christgen M, Kuemmel S, Grischke EM, Forstbauer H, Braun M, Warm M, Hackmann J, Uleer C, Aktas B, Schumacher C, Wuerstlein R, Pelz E, Kreipe HH, Clark SJ, Trau M, Graeser M, Harbeck N. Immunomodulatory gene networks predict treatment response and survival to de-escalated, anthracycline-free neoadjuvant chemotherapy in triple-negative breast cancer in the WSG-ADAPT-TN trial. Mol Cancer. 2025 Mar 26;24(1):96. doi: 10.1186/s12943-025-02275-0. PMID 40140821
- [Derived] Richters L, Gluz O, Weber-Lassalle N, Christgen M, Haverkamp H, Kuemmel S, Kayali M, Kates RE, Grischke EM, Altmuller J, Forstbauer H, Thiele H, Braun M, Warm M, Ossowski A, Wuerstlein R, Ernst C, Graeser M, Linn SC, Nitz U, Hauke J, Kreipe HH, Schmutzler RK, Hahnen E, Harbeck N. Genetic Alterations, Therapy Response, and Survival Among Patients With Triple-Negative Breast Cancer: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2025 Feb 3;8(2):e2461639. doi: 10.1001/jamanetworkopen.2024.61639. PMID 40009381
- [Derived] Kolberg-Liedtke C, Feuerhake F, Garke M, Christgen M, Kates R, Grischke EM, Forstbauer H, Braun M, Warm M, Hackmann J, Uleer C, Aktas B, Schumacher C, Kuemmel S, Wuerstlein R, Graeser M, Nitz U, Kreipe H, Gluz O, Harbeck N. Impact of stromal tumor-infiltrating lymphocytes (sTILs) on response to neoadjuvant chemotherapy in triple-negative early breast cancer in the WSG-ADAPT TN trial. Breast Cancer Res. 2022 Sep 2;24(1):58. doi: 10.1186/s13058-022-01552-w. PMID 36056374
- [Derived] Gluz O, Nitz U, Kolberg-Liedtke C, Prat A, Christgen M, Kuemmel S, Mohammadian MP, Gebauer D, Kates R, Pare L, Grischke EM, Forstbauer H, Braun M, Warm M, Hackmann J, Uleer C, Aktas B, Schumacher C, Wuerstlein R, Graeser M, Pelz E, Jozwiak K, Zu Eulenburg C, Kreipe HH, Harbeck N; ADAPT TN investigators. De-escalated Neoadjuvant Chemotherapy in Early Triple-Negative Breast Cancer (TNBC): Impact of Molecular Markers and Final Survival Analysis of the WSG-ADAPT-TN Trial. Clin Cancer Res. 2022 Nov 14;28(22):4995-5003. doi: 10.1158/1078-0432.CCR-22-0482. PMID 35797219
- [Derived] Graeser M, Schrading S, Gluz O, Strobel K, Herzog C, Umutlu L, Frydrychowicz A, Rjosk-Dendorfer D, Wurstlein R, Culemann R, Eulenburg C, Adams J, Nitzsche H, Prange A, Kummel S, Grischke EM, Forstbauer H, Braun M, Potenberg J, von Schumann R, Aktas B, Kolberg-Liedtke C, Harbeck N, Kuhl CK, Nitz U. Magnetic resonance imaging and ultrasound for prediction of residual tumor size in early breast cancer within the ADAPT subtrials. Breast Cancer Res. 2021 Mar 18;23(1):36. doi: 10.1186/s13058-021-01413-y. PMID 33736679